CLINICAL TRIAL: NCT02772809
Title: Usability Testing of Affordable Haptic Robots for Stroke Therapy
Acronym: Theradrive
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The robot was no longer available to the study.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 819787
Record Dates: First submitted 2016-03-29; First posted 2016-05-16 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Stroke; Hemiplegia
Keywords: stroke; hemiplegia; rehabilitation; robotics; neuroplasticity
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stroke survivors with low and moderate motor deficits (Other): Subjects with low and moderate motor deficits will 1) complete exercises with 2 commercial (joystick and wheel) and the Theradrive haptic robot after pre assessment 2) then experience 12 therapy sessions on the Theradrive haptic robot with Adaptive Feedback. 3) Assessments pre and post therapy.
  Interventions: Device: Haptic Robot Therapy with Games

INTERVENTIONS:
Device: Haptic Robot Therapy with Games — Commercial Joystick and Wheels Plus the Haptic TheraDrive Robot will be used. Haptic Theradrive is a low-cost robotic system for post-stroke upper extremity rehabilitation. The system uses off-the-shelf computer gaming wheels with force feedback to help reduce motor impairment and improve function in the arms of stroke survivors.

SUMMARY:
Stroke survivors with hemiplegia will be evaluated by rehabilitation professionals and asked to perform a battery of assessments to test the viability and usability of a force-feedback robot that adapts to each individual subject's performance. Subsequently, they will be asked to complete post-assessment questionnaires that provide feedback to the researchers on their observations and thoughts about the therapy devices.

DETAILED DESCRIPTION:
TheraDrive is a low-cost robotic system for post-stroke upper extremity rehabilitation. The system uses off-the-shelf computer gaming wheels with force feedback to help reduce motor impairment and improve function in the arms of stroke survivors. Preliminary results from various studies have shown that the original TheraDrive system lacked a robust mechanical linkage which could withstand the forces exerted by patients, lacked a patient-specific adaptive controller to deliver personalized therapy, and was not capable of delivering effective therapy to severely low-functioning patients. A new low-cost, high-force haptic robot with a single degree of freedom has been developed to address these concerns. This study has two purposes: first, to test the viability and usability of the new robot system alongside the original TheraDrive system; and second, to test if low-functioning patients benefit, and if so how much, from using force-feedback therapy as opposed to devices with zero impedance. This will be done by recruiting approximately 36 human subjects. Exercises will be performed by study subjects and an adaptive controller will monitor patient performance to ensure that exercises are difficult but doable, which is important for maintaining patient motivation. It is hypothesized that not only will the new system be viable, but that it will provide better robot-assisted therapy to a large variety of patients, especially low-functioning stroke survivors with hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors at least 18 years of age with hemiplegia.
* The subject's stroke must have occurred at least 3 months prior to enrollment in the study.
* Low and Moderate functioning stroke survivors as measured by Fugl- Meyer
* Not depressed
* No more than Mild Cognitive Deficit
* Participants must be able to sit upright for 4 hours at a time in Part A of the study; and 2 hours at a time, 3 days a week, for Part B of the study.
* The subject's stroke must have occurred at least 3 months prior to enrollment in the study.

Exclusion Criteria:

* Greater than mild cognitive deficits
* Greater than mild depression. A member of the research team will administer Beck's Depression Inventory (BDI) to each study participant over the phone. If the participant is found to have greater than mild depression, as measured by the BDI, they will not qualify for the study.
* Receiving rehabilitation on the upper limb.
* Received Botox injections within the past 3 months.
* Suffering from contractures (chronic loss of joint motion) or debilitating spasticity in the upper extremity.
* Experiencing greater than mild pain, and/or the PI determines that the participant should no longer continue working with the novel therapy devices, the study will be stopped.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Johnson, PhD, Principal Investigator — PENN MEDICINE RITTENHOUSE
Locations (1):
- Penn Medicine Rittenhouse, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruparel R, Johnson MJ, Strachota E, McGuire J, Tchekanov G. Evaluation of the TheraDrive system for robot/computer assisted motivating rehabilitation after stroke. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:811-4. doi: 10.1109/IEMBS.2009.5332386. PMID 19963475
- [Background] Johnson MJ, Ramachandran B, Paranjape RP, Kosasih JB. Feasibility study of TheraDrive: a low-cost game-based environment for the delivery of upper arm stroke therapy. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:695-8. doi: 10.1109/IEMBS.2006.259971. PMID 17946851
- [Background] Theriault A, Nagurka M, Johnson MJ. Design and development of an affordable haptic robot with force-feedback and compliant actuation to improve therapy for patients with severe hemiparesis. IEEE Trans Haptics. 2014 Apr-Jun;7(2):161-74. doi: 10.1109/TOH.2013.51. PMID 24968380
- See also: A computer model of the human arm: Predictive biomechanics for the theradrive rehabilitation system — https://doi.org/10.1109/ICORR.2015.7281300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stroke survivors over the age of 18 with hemiplegia, who are three months post event, and have varying levels of impairment in the upper extremities will be recruited. All use of the TheraDrive system will take place at the Rehabilitation Robotics Lab on the ﬁrst ﬂoor of Penn Rittenhouse
Groups:
- Stroke Survivors With Varying Levels of Motor Impairment: Stroke survivors with varying levels of motor deﬁcit impairment in their upper extremity.
Period: Overall Study
Arm/Group | Stroke Survivors With Varying Levels of Motor Impairment
Started | 23
Completed | 17
Not Completed | 6
Not completed — not completed some tasks | 6

BASELINE CHARACTERISTICS:
Population: Severe motor deficit participants were not included in this study.
Groups:
- Subjects With Varying Levels of Motor Impairment: Subjects with varying levels of motor impairments who are ages 18 and older.
Arm/Group | Subjects With Varying Levels of Motor Impairment
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 6 persons did not complete all of the tracking tasks so the data was excluded.
  Participants
    number analyzed (Participants) | 17
    Female | 9
    Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Fugl Meyer
Description: The primary outcomes are motor control for the upper limb: Subjects completed tasks on scale; Motor scale maximum is 66. minimum is 0. Lower is more impaired. Higher is less impaired.
Time Frame: At 0 weeks
Population: 6 subjects did not complete so not included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stroke Survivors With Motor Impairment: All subject used robot for tracking tasks
Arm/Group | Stroke Survivors With Motor Impairment
Number analyzed (Participants) | 17
score on a scale | 42.5 (20.2)

2. Primary Outcome: Box and Blocks
Description: Measures ADL Function. Completed reach and grasp activities. Reached for 1 inch cube and placed with impaired arm. More blocks indicate higher function. Less blocks lower function
Time Frame: At Session 0. Pre-intervention
Population: 6 subjects did not complete so not included in the analysis
Measure: Mean (Standard Deviation); unit: # of blocks
Groups:
- Subjects With Motor Impairment: Subjects with deﬁcit ages 18 and older.
Arm/Group | Subjects With Motor Impairment
Number analyzed (Participants) | 17
# of blocks | 19.11 (15.49)

3. Primary Outcome: Tracking Accuracy
Description: Tracking accuracy is measured using the normalized root mean square, which is a measure for error in tracking performance with respect to a desired goal. Root mean squared divided by the maximum error if person does not move. The higher the decimal the higher the error made. Lower is better performance.
Time Frame: At Session 0
Population: 6 subjects did not complete so not included in the analysis
Measure: Mean (Standard Deviation); unit: accuracy index
Groups:
- Stroke Survivors With Motor Impairments: All subject used robot for tracking tasks
Arm/Group | Stroke Survivors With Motor Impairments
Number analyzed (Participants) | 17
accuracy index | 0.73 (0.44)

4. Secondary Outcome: Grip Strength
Description: Grip strength as measured by a dynamometer. Subjects were asked to squeeze a dynamometer with impaired arm. Higher forces mean better function
Time Frame: pre-intervention
Population: 6 subjects did not complete so not included in the analysis
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- Subjects With Motor Impairment: Subjects completed tasks with robot and with clinical scale.
Arm/Group | Subjects With Motor Impairment
Number analyzed (Participants) | 17
lbs | 26.88 (22.73)

5. Secondary Outcome: Montreal Cognitive Assessment (MOCA)
Description: A brief 30-question test that takes around 10 to 12 minutes to complete and helps assess people for impairment in cognition domains. Maximum is 30. Minimum is 0; Low is <17 is severe cognitive impairment; a score 26 and higher is normal cognition.
Time Frame: pre-intervention
Population: 6 subjects did not complete so not included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Subjects With Motor Impairments: Subjects with motor impairments who are ages 18 and older.
Arm/Group | Subjects With Motor Impairments
Number analyzed (Participants) | 17
units on a scale | 22.5 (4.6)

6. Secondary Outcome: Becks Depression Scale
Description: Measures depression. The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression (Beck, et al., 1961). Maximum is 63 Total Score_______________Levels of Depression 1-10____________________These ups and downs are considered normal 11-16___________________ Mild mood disturbance 17-20___________________Borderline clinical depression 21-30___________________Moderate depression 31-40___________________Severe depression over 40__________________Extreme depression
Time Frame: Pre-intervention
Population: 6 subjects did not complete so not included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stroke Survivors With Motor Impairments: All subject used robot for tracking tasks;
Arm/Group | Stroke Survivors With Motor Impairments
Number analyzed (Participants) | 17
units on a scale | 7.25 (5.72)

ADVERSE EVENTS:
Time Frame: 40 months
Description: No adverse events were reported.
Groups:
- Haptic Robot Therapy With Games: Subjects with low and moderate motor deficits will 1) complete exercises with 2 commercial (joystick and wheel) and the Theradrive haptic robot after pre assessment 2) then experience 12 therapy sessions on the Theradrive haptic robot with Adaptive Feedback. 3) Assessments pre and post therapy.
  Haptic Robot Therapy with Games: Commercial Joystick and Wheels Plus the Haptic TheraDrive Robot will be used. Haptic Theradrive is a low-cost robotic system for post-stroke upper extremity rehabilitation. The system uses off-the-shelf computer gaming wheels with force feedback to help reduce motor impairment and improve function in the arms of stroke survivors.
Arm/Group | Haptic Robot Therapy With Games
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT02772809/Prot_SAP_000.pdf